CLINICAL TRIAL: NCT06925152
Title: COMFORT Trial: Complex Obstetric Management With Focused Regional Transversus Abdominis Plane Block
Acronym: COMFORT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Regional One Health (Other)
Responsible Party: Principal Investigator, Michael B VanDillen MD, Principal Investigator, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMFORT2025
Record Dates: First submitted 2025-03-19; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Complex Obstetric Surgery; Perioperative Pain Management; Cesarean Delivery; Postoperative Pain Control
Keywords: Complex obstetric surgery; Perioperative pain management; cesarean delivery; postoperative pain control

STUDY DESIGN:
Intervention Model Description: Multi-year (February 2025- February 2028) prospective double blinded randomized-control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators plan to perform a double-blind study. Other than the investigational pharmacists, who do not have direct participant interaction, all study investigators and clinical care providers will be blinded to the allocation of participants. All clinical care will be per standard protocols for all participants. Patients will be unaware of their assignment. Data collectors/outcomes assessors will similarly collect all data and outcomes unaware of the assignment. All interim safety analyses and reports to the Data Safety Monitoring board will be blinded, with groups reported as A and B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator): Placebo group TAP (Transversus Abdominis Plane) block syringe will include 30mL normal saline.
  Interventions: Drug: Placebo arm
- Intervention group (Active Comparator): TAP (Transversus Abdominis Plane) blocks will include 0.5% bupivacaine in 30mL solution of 15mL normal saline and 15mL bupivacaine.
  Interventions: Drug: Bupivicaine intervention arm

INTERVENTIONS:
Drug: Bupivicaine intervention arm — TAP blocks in intervention group will include 0.5% bupivacaine in 30mL solution of 15mL normal saline and 15mL bupivacaine
  Arms: Intervention group
Drug: Placebo arm — Placebo group TAP block syringe will include 30mL normal saline
  Arms: Placebo group

SUMMARY:
To assess the effect of intraoperative transversus abdominis plane (TAP) blocks on the amount of opioid pain medications expressed as morphine milliequivalents (MME) used postoperatively in patients who have undergone cesarean delivery (CD) in the setting of complex obstetric surgery (COS).

DETAILED DESCRIPTION:
The Transversus Abdominis Plane (TAP) block is a regional anesthesia technique that targets the nerves innervating the abdominal wall, providing effective postoperative analgesia for patients undergoing various abdominal surgeries, including cesarean deliveries. The standard clinical practice for TAP blocks typically involves local anesthetics like bupivacaine, which, when administered in the appropriate plane, has been shown to reduce opioid consumption and improve pain management in the postoperative period.

Transversus abdominal plane (TAP) blocks, when administered intraoperatively, have demonstrated significant benefits in managing postoperative pain, especially in abdominal surgeries. Placing the TAP block during surgery provides early and prolonged analgesia, potentially reducing the need for postoperative opioids and improving recovery outcomes. A study completed in 2007 was one of the first to highlight the effectiveness of intraoperative TAP block placement in patients undergoing lower abdominal surgeries, showing a significant reduction in opioid consumption and better pain control. In the context of cesarean section, an intraoperative TAP block was shown to provide effective analgesia with a reduction in postoperative narcotic use. Similarly, a randomized trial in 2017 demonstrated that intraoperative TAP blocks significantly improved pain scores and reduced opioid consumption in patients undergoing colorectal surgeries. Furthermore, a study completed in 2014 found that performing TAP blocks intraoperatively for laparoscopic cholecystectomy patients resulted in lower visual analog scale (VAS) pain scores in the recovery room and reduced the incidence of postoperative nausea and vomiting. These findings underscore the advantages of intraoperative TAP block placement in enhancing postoperative analgesia across a variety of abdominal procedures.

Despite the widespread use of TAP blocks, there remains a gap in the literature regarding the effectiveness of bupivacaine TAP block use placed intraoperatively during more complex obstetric surgeries. Most existing studies focus on the use of TAP blocks for pain management after routine Pfannenstiel cesarean deliveries, with limited attention given to their role in cases involving higher-risk or more complicated obstetric situations, such as cesareans with significant intra-abdominal adhesions or other complications.

Although bupivacaine is commonly used in TAP blocks, its specific efficacy, optimal dosing, and potential benefits when placed intraoperatively in complex obstetric cases remain underexplored. The limited data in this area presents a critical gap in our understanding of how best to optimize pain management and improve surgical outcomes for women undergoing cesarean delivery, particularly in high-risk obstetric cases.

This blinded randomized controlled trial (RCT) seeks to address this gap by evaluating the effectiveness of intraoperative TAP blocks with bupivacaine during complex cesarean sections, focusing on the impact on postoperative analgesia and pain scores. By clarifying the role of bupivacaine in TAP blocks during complex obstetric surgery, this study aims to contribute valuable insights to the field of obstetric anesthesia and improve the perioperative experience for patients undergoing cesarean delivery.

Primary Objective: To assess the effect of intraoperative transversus abdominis plane (TAP) blocks on the amount of opioid pain medications expressed as morphine milliequivalents (MME) used postoperatively in patients who have undergone cesarean delivery (CD) in the setting of complex obstetric surgery (COS).

Primary Endpoint/Outcome: Pain medication requested, expressed as MMEs, between 24 and 48 hours after surgery.

Secondary Endpoint(s)/Outcome(s):

Total MME requested within first 24-hours post operatively Total MME requested within 48-hours post operatively Total MME at 1-week after surgery Functional assessment of activities of daily life (ADL) at 1-week post operatively Number of unplanned postoperative visits within 6-months of surgery Geographic region of patients needing complex obstetric surgery. Heat maps: diversity equity and inclusion (DEI) zip codes

Hypothesis: The investigators hypothesize that utilization of the TAP block will reduce MME requirements by 20% for patients who have undergone CD in the setting of COS.

ELIGIBILITY:
Inclusion criteria:

Patient has a history of a least one of the following:

* Prior exploratory laparotomy
* History of non-obstetric open intra-abdominal surgery
* History of three or more prior cesarean deliveries
* History of intra-abdominal or pelvic adhesive disease
* History of abdominoplasty
* History of abdominal re-exploration surgery

Exclusion Criteria:

* Received general anesthesia
* History of less than 3 cesarean deliveries if do not meet other inclusion criteria
* History of chronic opioid use
* History of substance abuse (i.e. alcohol, methamphetamine/amphetamine, abuse of prescription opioid medication, or heroin use)
* History of chronic kidney disease
* Allergies to bupivacaine or oral analgesics
* Patient preference
* Cesarean hysterectomy
* Administration of ≥4mg morphine to epidural
* Loss to follow-up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Pain medication requested | Between 24 and 48 hours after surgery
  Total pain medication requested expressed in morphine milligram equivalents.

SECONDARY OUTCOMES:
Total MME requested within first 24 hours postoperatively | 24 hours postoperatively
Total MME requested within 48 hours postoperatively | 48 hours postoperatively
Total MME at one week after surgery | One week postoperatively
Functional assessment of activities of daily life (ADL) at one week postoperatively | One week postoperatively
Number of unplanned postoperative visits within six months of surgery | Six months postoperatively
Geographic region of patients needing complex obstetric surgery | 24 months - through the duration of the study
  Heat maps to evaluate the distribution of patients across different demographic categories based on race and age within certain zip codes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Johns N, O'Neill S, Ventham NT, Barron F, Brady RR, Daniel T. Clinical effectiveness of transversus abdominis plane (TAP) block in abdominal surgery: a systematic review and meta-analysis. Colorectal Dis. 2012 Oct;14(10):e635-42. doi: 10.1111/j.1463-1318.2012.03104.x. PMID 22632762
- [Background] Zhang, X., et al. (2017).
- [Background] Kehlet, H., et al. (2014).
- [Background] Garmi G, Parasol M, Zafran N, Rudin M, Romano S, Salim R. Efficacy of Single Wound Infiltration With Bupivacaine and Adrenaline During Cesarean Delivery for Reduction of Postoperative Pain: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2242203. doi: 10.1001/jamanetworkopen.2022.42203. PMID 36378307
- [Background] Abdallah FW, Halpern SH, Margarido CB. Transversus abdominis plane block for postoperative analgesia after Caesarean delivery performed under spinal anaesthesia? A systematic review and meta-analysis. Br J Anaesth. 2012 Nov;109(5):679-87. doi: 10.1093/bja/aes279. Epub 2012 Aug 19. PMID 22907337
- [Background] Ueshima, H., Higashijima, U., Matsumoto, M., & Imai, S. (2013). The effect of the volume of local anesthetic on the analgesic effect of transversus abdominis plane block in abdominal surgery. Journal of Anesthesia, 27(6), 650-655.